CLINICAL TRIAL: NCT01177956
Title: Open-label, Single-arm, Multicenter, Phase III Trial to Assess the Antitumor Activity and Safety Profile of Cetuximab When Given in Combination With Chemotherapy for the First-line Treatment of Recurrent and/or Metastatic Squamous Cell Carcinoma of the Head and Neck in Asian Subjects
Brief Title: A Trial to Determine the Safety and Anti-tumor Activity Profile of the Combination of Cetuximab and Concomitant Cisplatin Plus 5-Fluorouracil (5-FU) in Subjects With Recurrent and/or Metastatic Squamous Cell Carcinoma in Head and Neck
Acronym: CHANGE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR62241_055
Record Dates: First submitted 2010-06-02; First posted 2010-08-09 (Estimated); Results first posted 2012-08-10 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-08

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: Recurrent and/or metastatic squamous cell carcinoma of the head and neck; 1st-line; Cetuximab; Chemotherapy; EMR 62241 -055; Merck KGaA; Recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab + Cisplatin + 5-Fluorouracil (5-FU) (Experimental)
  Interventions: Biological: Cetuximab; Drug: Cisplatin; Drug: 5-Fluorouracil

INTERVENTIONS:
Biological: Cetuximab — The initial dose of cetuximab will be 400 milligram per square meter (mg/m^2) as an intravenous (IV) infusion over 120 minutes. Subsequent weekly doses will be 250 mg/m^2 as an IV infusion over 60 minutes.
  Chemotherapy will be continued for up to a maximum of six 3-week cycles in the absence of progressive disease (PD) or unacceptable toxicity. All subjects will receive cetuximab treatment until the occurrence of PD or unacceptable toxicity to cetuximab.
  Other Names: Erbitux®
Drug: Cisplatin — Subjects will receive 75 mg/m^2 cisplatin as an IV infusion over 60 minutes on day 1 of each 3-week treatment cycle.
Drug: 5-Fluorouracil — Subjects will receive 750 mg/m^2 per day 5-FU as a continuous IV infusion over 24 hours from day 1 to day 5 of each 3-week treatment cycle.

SUMMARY:
The primary objective of this trial is to assess the antitumor activity and safety profile of cetuximab when given in combination with cisplatin + 5-Fluorouracil (5-FU) for the first-line treatment of recurrent and/or metastatic Squamous Cell Carcinoma in Head and Neck (SCCHN) in Asian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Inpatient
* Greater than or equal to (>=) 18 years of age
* Histologically or cytologically confirmed diagnosis of SCCHN
* Recurrent and/or metastatic SCCHN not suitable for local therapy
* Presence of at least 1 measurable lesion identified either by computed tomography (CT) scan or magnetic resonance imaging (MRI) according to modified WHO criteria
* Karnofsky performance status (KPS) >= 80 percent at trial entry
* Neutrophils >= 1.5*10^9 per liter (L), platelet count >= 100*10^9 per L, and hemoglobin >= 90 gram per liter (g/L)
* Total bilirubin less than or equal to (<=) 2*upper limit of normal (ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=3*ULN
* Serum creatinine <=133 micromole per liter (mcmol/L)
* Serum calcium within normal range
* Effective contraception if procreative potential exists (applicable for both male and female subjects)

Exclusion Criteria:

* Prior systemic chemotherapy, except if given as part of a multimodal treatment which was completed more than 6 months prior to trial entry
* Surgery (excluding prior diagnostic biopsy) or irradiation within 4 weeks before trial entry
* Nasopharyngeal carcinoma
* Active infection (infection requiring IV antibiotics), including active tuberculosis, or known and declared human immunodeficiency virus (HIV)
* Uncontrolled diabetes mellitus, pulmonary fibrosis, acute pulmonary disorder, interstitial pneumonia, cardiac failure or liver failure
* Uncontrolled hypertension defined as systolic blood pressure >=180 millimeter of mercury (mmHg) and/or diastolic blood pressure >=130 mmHg under resting conditions
* Pregnancy (absence to be confirmed by serum beta human chorionic gonadotrophin [beta-HCG] test) or breastfeeding
* Concomitant chronic systemic immune therapy or hormonal therapy as cancer therapy
* Other concomitant anticancer therapies
* Documented or symptomatic brain or leptomeningeal metastasis
* Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months or high risk of uncontrolled arrhythmia or uncontrolled cardiac insufficiency
* Medical or psychological condition that would not permit the subject to complete the trial or sign informed consent
* Known drug abuse (with the exception of alcohol abuse)
* Known hypersensitivity or allergic reaction against any of the components of the trial treatment
* Previous treatment with monoclonal antibody therapy, other signal transduction inhibitors or epidermal growth factor receptor (EGFR) targeting therapy
* Previous or current other squamous cell carcinoma (SCC)
* Evidence of previous other malignancy within the last 5 years
* Signs and symptoms suggestive of transmissible spongiform encephalopathy, or family members who suffer(ed) from such
* Intake of any investigational medication within 30 days before trial entry
* Legal incapacity or limited legal capacity
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-12; Primary Completion 2011-01 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- China (13):
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing
  - Jilin Cancer Hospital, Changchun
  - The Xiangya 2nd Hospital of Central South University, Changsha
  - Fuijan Provincial Tumor Hospital, Fuijian
  - Nanfang Hospital of Nanfang Medical University, Guangzhou
  - Sun Yat-Sen Univesity Cancer Center, Guangzhou
  - Zhejiang Provincial Tumor Hospital, Hangzhou
  - Jiangsu Cancer Hospital, Jiangsu, Nanjing
  - Tumor Hospital of Guangxi Zhuang Autonomous Region / The Tumor Affiliated Hospital of Guangxi Medical University, Nanning
  - Eye & ENT Hospital of Fundan University, Shanghai
  - Fundan University Shanghai Cancer Center, Shanghai
  - Tongji Hospital of Tongji Medical College of Huazhong University of Science & Technology, Wuhan
  - Xijing Hospital, the Fourth Military Medical University, Xi'an
- Clinical Trial Center of Medical Research Institute, Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Result] Guo Y, Shi M, Yang A, Feng J, Zhu X, Choi YJ, Hu G, Pan J, Hu C, Luo R, Zhang Y, Zhou L, Cheng Y, Lupfert C, Cai J, Shi Y. Platinum-based chemotherapy plus cetuximab first-line for Asian patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck: Results of an open-label, single-arm, multicenter trial. Head Neck. 2015 Aug;37(8):1081-7. doi: 10.1002/hed.23707. Epub 2014 Sep 17. PMID 24710768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last participant (informed consent): December 2009/September 2010. Clinical data cut-off: 25 January 2011, Study completion date: November 2012
Pre-assignment Details: A total of 73 participants were enrolled, out of which 5 participants were screen failure and 68 participants received the study treatment.
Groups:
- Cetuximab + Cisplatin + 5-FU: Participants were administered an initial dose of cetuximab 400 milligram per square meter (mg/m^2) intravenous (IV) infusion over 120 minutes followed by subsequent weekly doses of 250 mg/m^2 IV infusion over 60 minutes along with background chemotherapy consisting of cisplatin 75 mg/m^2 IV infusion over 60 minutes on day 1 of each 3-week treatment cycle and 5-fluorouracil (5-FU) 750 mg/m^2 per day as a continuous IV infusion over 24 hours from day 1 to day 5 of each 3-week treatment cycle, for up to 6 cycles in the absence of progressive disease (PD) or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cetuximab + Cisplatin + 5-FU
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population included all participants who received at least one dose of the investigational medicinal product (IMP) cetuximab or chemotherapy.
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (9.5)
Age, Customized [Number; unit: participants]
  <65 years | 55
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 49
Race/Ethnicity, Customized [Number; unit: participants]
  Asian (Chinese) | 63
  Asian (Korean) | 5

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) Until Cut-off Date 25 January 2011
Description: BOR: Percentage of participants experiencing a Complete Response (CR) (complete disappearance of measurable and evaluable disease without new lesions) or Partial Response (PR) (greater than or equal to 50 percent decrease of sum of product diameters of measurable disease, evaluable disease not worsening or progressing, no new lesions confirmed by a subsequent assessment no less than 28 days after criteria for response were first met) (based on modified World Health Organization [WHO] criteria), divided by the number of participants belonging to intention to treat (ITT) or safety population.
Time Frame: Evaluations were performed every 6 weeks until progression, reported between day of first participant randomized, 25 December 2009, until cut-off date 25 January 2011
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
percentage of participants | 54.4 [41.9 to 66.5]

2. Secondary Outcome: Overall Survival (OS) Time Until Cut-off Date 15 November 2012
Description: The OS time was defined as the time from first administration of trial treatment to death. Participants without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized, 25 December 2009, until cut-off date 15 November 2012
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
months | 12.6 [9.1 to 15.0]

3. Secondary Outcome: Progression-free Survival (PFS) Time Until Cut-off Date 25 January 2011
Description: Duration from first administration of trial treatment until progression (radiological or clinical, if radiological progression is not available) or death due to any cause. Only deaths within 60 days of last tumor assessment are considered. Participants without event are censored on the date of last tumor assessment.
Time Frame: as for outcome 1
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
months | 6.2 [5.1 to 8.1]

4. Secondary Outcome: Progression-free Survival (PFS) Time Until Cut-off Date 15 November 2012
Description: as for outcome 3
Time Frame: Evaluations were performed every 6 weeks until progression, reported between day of first participant randomized, 25 December 2009, until cut-off date 15 November 2012
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
months | 6.6 [5.1 to 7.7]

5. Secondary Outcome: Time to Progression (TTP) Until Cut-off Date 25 January 2011
Description: Time from first administration of trial treatment to disease progression (radiological or clinical, if radiological progression is not available). Participants without event are censored on the date of last tumor assessment.
Time Frame: as for outcome 1
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
months | 6.8 [5.3 to 8.1]

6. Primary Outcome: Best Overall Response (BOR) Until Cut-off Date 15 November 2012
Description: BOR: Percentage of participants experiencing a CR (complete disappearance of measurable and evaluable disease without new lesions) or PR (greater than or equal to 50 percent decrease of sum of product diameters of measurable disease, evaluable disease not worsening or progressing, no new lesions confirmed by a subsequent assessment no less than 28 days after criteria for response were first met) (based on modified WHO criteria), divided by the number of participants belonging to ITT or safety population.
Time Frame: as for outcome 4
Population: ITT population included all participants who received at least one dose of the investigational medicinal product (IMP) cetuximab or chemotherapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
percentage of participants | 55.9 [43.3 to 67.9]

7. Secondary Outcome: Time to Progression (TTP) Until Cut-off Date 15 November 2012
Description: as for outcome 5
Time Frame: as for outcome 4
Population: ITT population included all participants who received at least one dose of the IMP cetuximab or chemotherapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 68
months | 7.0 [5.6 to 8.1]

8. Secondary Outcome: Duration of Response Until Cut-off Date 25 January 2011
Description: Time from first assessment of CR or PR to disease progression or death (within 60 days of last tumor assessment). Participants without event are censored on the date of last tumor assessment. Tumor assessments based on modified WHO criteria.
Time Frame: as for outcome 1
Population: Subgroup of participants from the study population having best confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 37
months | 5.7 [4.2 to 9.1]

9. Secondary Outcome: Duration of Response Until Cut-off Date 15 November 2012
Description: as for outcome 8
Time Frame: as for outcome 4
Population: Subgroup of participants from the study population having best confirmed response (CR or PR).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab + Cisplatin + 5-FU
Number analyzed (Participants) | 38
months | 6.1 [5.4 to 7.8]

ADVERSE EVENTS:
Time Frame: Baseline until 30 days after last trial treatment
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an IMP regardless of causal relationship and even if no IMP has been administered.
Groups:
- Cetuximab + Cisplatin + 5-FU : Treatment Emergent Phase: Participants were administered an initial dose of cetuximab 400 milligram per square meter (mg/m^2) intravenous (IV) infusion over 120 minutes followed by subsequent weekly doses of 250 mg/m^2 IV infusion over 60 minutes along with background chemotherapy consisting of cisplatin 75 mg/m^2 IV infusion over 60 minutes on day 1 of each 3-week treatment cycle and 5-fluorouracil (5-FU) 750 mg/m^2 per day as a continuous IV infusion over 24 hours from day 1 to day 5 of each 3-week treatment cycle, for up to 6 cycles in the absence of progressive disease (PD) or unacceptable toxicity. On or after the first dosing day of trial treatment and until 30 days after the last trial treatment administration.
- Cetuximab + Cisplatin + 5-FU : Late Phase: Participants were administered an initial dose of cetuximab 400 milligram per square meter (mg/m^2) intravenous (IV) infusion over 120 minutes followed by subsequent weekly doses of 250 mg/m^2 IV infusion over 60 minutes along with background chemotherapy consisting of cisplatin 75 mg/m^2 IV infusion over 60 minutes on day 1 of each 3-week treatment cycle and 5-fluorouracil (5-FU) 750 mg/m^2 per day as a continuous IV infusion over 24 hours from day 1 to day 5 of each 3-week treatment cycle, for up to 6 cycles in the absence of progressive disease (PD) or unacceptable toxicity. Participants with end of treatment date after the last trial treatment date + 30 days or still on trial at the cut-off date.
Arm/Group | Cetuximab + Cisplatin + 5-FU : Treatment Emergent Phase | Cetuximab + Cisplatin + 5-FU : Late Phase
Serious Adverse Events (participants affected / at risk) | 13/68 | 0/32
Other Adverse Events (participants affected / at risk) | 67/68 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Cisplatin + 5-FU : Treatment Emergent Phase (N=68) | Cetuximab + Cisplatin + 5-FU : Late Phase (N=32)
Anaphylactic reaction (Immune system disorders) | 2 (3) | 0 (0)
Microcytic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Mouth hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab + Cisplatin + 5-FU : Treatment Emergent Phase (N=68) | Cetuximab + Cisplatin + 5-FU : Late Phase (N=32)
Leucopenia (Blood and lymphatic system disorders) | 29 (98) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 19 (42) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (9) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (9) | 0 (0)
Constipation (Gastrointestinal disorders) | 21 (35) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (17) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 8 (11) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (59) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 4 (4) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 12 (32) | 0 (0)
Vomiting (Gastrointestinal disorders) | 19 (48) | 0 (0)
Asthenia (General disorders) | 7 (12) | 0 (0)
Fatigue (General disorders) | 10 (21) | 0 (0)
Mucosal Inflammation (General disorders) | 9 (17) | 0 (0)
Pyrexia (General disorders) | 15 (20) | 0 (0)
Paronychia (Infections and infestations) | 5 (5) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 5 (5) | 0 (0)
Hemoglobin Decreased (Investigations) | 13 (24) | 0 (0)
Neutrophil Count Decreased (Investigations) | 9 (14) | 0 (0)
Weight Decreased (Investigations) | 29 (38) | 0 (0)
Weight Increased (Investigations) | 5 (8) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 6 (18) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 18 (35) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Hypochloremia (Metabolism and nutrition disorders) | 5 (7) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 22 (43) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 (37) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 13 (23) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 0 (0)
Dizziness (Nervous system disorders) | 6 (8) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (8) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 13 (14) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (15) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 24 (46) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All submissions by the PI for publication require the written permission from the sponsor. The PI commits to forward to the sponsor all documents intended for publication which contains data or results generated in connection with the study. Documents must be available at least 60 days before the planned submission date to allow for review. Any publication should follow the policy in the protocol. The PI shall not publish results derived from the study until the study has been reported in full.